CLINICAL TRIAL: NCT03735537
Title: Treatment of Osteogenesis Imperfecta With Parathyroid Hormone and Zoledronic Acid
Acronym: TOPaZ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC16092; 2016-003228-22 (EudraCT Number)
Record Dates: First submitted 2018-08-09; First posted 2018-11-08 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Osteogenesis Imperfecta
Keywords: Fracture; Teriparatide
MeSH Terms: conditions — Osteogenesis Imperfecta; Fractures, Bone | interventions — Teriparatide; Zoledronic Acid; Solutions

STUDY DESIGN:
Intervention Model Description: Multicentre, parallel arm, open-label, phase IV randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: Images of incident fractures and vertebral fractures will be assessed by an independent clinical adjudicator blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teriparatide and zoledronic acid (Active Comparator): Teriparatide (TPTD) 20mcg daily using Teriparatide Pen Injector, given subcutaneously using a self-administered injection device for two years (24 months) followed by a single intravenous 5mg infusion of zoledronic acid.
  Interventions: Drug: Teriparatide Pen Injector; Drug: Zoledronic Acid
- Standard Care (No Intervention): Continuation of existing bone modifying treatment (i.e. bisphosphonate treatment) or no active bone modifying treatment according to the clinical judgement of the local investigator.

INTERVENTIONS:
Drug: Teriparatide Pen Injector
  Other Names: Forsteo; Forteo
  Arms: Teriparatide and zoledronic acid
Drug: Zoledronic Acid — Any brand or preparation may be used to deliver the required dose of 5mg
  Other Names: Aclasta 5mg solution for infusion; Zoledronic acid 5mg/100ml solution for infusion
  Arms: Teriparatide and zoledronic acid

SUMMARY:
Osteogenesis imperfecta (OI) is an inherited skeletal disorder characterised by increased risk of fragility fractures. Bisphosphonates are frequently prescribed for adult patients with OI with the aim of preventing fractures but the evidence base for efficacy is poor. Recent evidence suggests that the bone anabolic agent teriparatide (TPTD) increases bone mineral density (BMD) and may have the potential to prevent fractures in OI.

The purpose of the TOPaZ Trial is to investigate if a a two-year course of teriparatide (TPTD) followed by antiresorptive therapy with a single infusion of zoledronic acid (ZA) in adults with OI reduces the proportion of patients who experience a fracture as compared with standard care

Adult patients with a clinical diagnosis of OI who are willing and able to give informed consent and who do not have contraindications to the study medications will be recruited from participating sites. Participants will be randomised 1:1 to receive either standard care for the duration of the trial or TPTD for 24 months followed by a single infusion of ZA, or another antiresorptive agent in the event that ZA is contraindicated.

Participants will attend recruiting centres for a Baseline/Screening visit, at 12 months, 24 months and at the end of the trial for formal study visits with telephone calls every 6 months from a site research nurse. Participants randomised to TPTD will also attend recruiting centre at regular intervals during the 24 month treatment period to collect new supplies of TPTD.

DETAILED DESCRIPTION:
Osteogenesis imperfecta (OI) is an inherited skeletal disorder characterised by increased risk of fragility fractures. Bisphosphonates are frequently prescribed for adult patients with OI with the aim of preventing fractures but the evidence base for efficacy is poor. Recent evidence suggests that the bone anabolic agent teriparatide (TPTD) increases bone mineral density (BMD) and may have the potential to prevent fractures in OI.

The purpose of the TOPaZ Trial is to investigate if a a two-year course of teriparatide (TPTD) followed by antiresorptive therapy with a single infusion of zoledronic acid (ZA) in adults with OI reduces the proportion of patients who experience a fracture as compared with standard care.

The trial has a number of secondary objectives which aim to investigate if a two-year course of TPTD followed by antiresorptive therapy with a single infusion of ZA in adults with OI reduces the total number of fractures, reduces the risk of vertebral fractures; or affects bone pain, quality of life and functional status as compared with standard care. There is also a planned mechanistic analysis to understand which baseline characteristics of adults with OI, such as age, clinical subtype of OI, genetic diagnosis, bone turnover, BMD, and previous treatment influences the occurrence of fractures and/or the response to treatment

Adult patients with a clinical diagnosis of OI who are willing and able to give informed consent and who do not have contraindications to the study medications will be recruited from participating sites. Participants will be randomised 1:1 to receive either standard care for the duration of the trial or TPTD for 24 months followed by a single infusion of ZA, or another antiresorptive agent in the event that ZA is contraindicated. Exclusion criteria include: current or previous treatment with an investigational (non-licensed experimental) drug with effects on bone metabolism, contraindication to TPTD or ZA, women of childbearing potential not using highly effective methods of contraception, pregnancy, women that are breastfeeding or age <18 years.

Participants will attend recruiting centres for a Baseline/Screening visit, at 12 months, 24 months and at the end of the trial for formal study visits with telephone calls every 6 months from a site research nurse. Participants randomised to TPTD will also attend recruiting centre at regular intervals during the 24 month treatment period to collect new supplies of TPTD.

The baseline assessment will include dual energy x-ray absorptiometry (DEXA), spine x-rays, safety bloods, medical and fracture history, pain (brief pain inventory, BPI) and quality of life (SF36, HAQ, EQ5D, PSQI). Blood will be taken for genetic analysis and for analysis of biochemical markers of bone turnover. In some centres, a high resolution quantitative CT scan (HRQCT) of the wrist and tibia will be performed. Participants will be seen after 12 months when bloods, questionnaires and HRQTC will be repeated; at 24 months when bloods, questionnaires, DEXA and HRQCT will be repeated. At the end of the study participants will undergo DEXA, spine x-rays, HRQCT and bloods and questionnaires will be repeated. Information on adverse events and fractures will be collected throughout the study and participants suspected to have fractures will have x-ray or other imaging to confirm the presence of fractures.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years and over with a clinical diagnosis of Osteogenesis Imperfecta (OI)
* Patients willing and able to consent and comply with the study protocol

Exclusion Criteria:

* Current or previous treatment with an investigational (non-licensed experimental) drug with effects on bone metabolism
* Contraindication to teriparatide or zoledronic acid
* Women of childbearing potential not using highly effective methods of contraception
* Pregnancy
* Women that are breastfeeding
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Incident clinical fractures validated by x-ray or other imaging | Through study completion, approximately 5 years
  Proportion of participants experiencing a clinical fracture validated by x-ray or other imaging as compared to standard care

SECONDARY OUTCOMES:
Total number of incident vertebral fractures | Baseline (0) and Final Trial Visit (5 years after baseline)
  Incident vertebral fractures assessed by imaging of the thoracic and lumbar spine and reviewed by an independent masked adjudicator using two spine x-rays collected at the start and end of the trial
Total number of fractures | Through study completion, approximately 5 years
  Total number of fractures experienced by participant defined as combination of validated clinical fractures, vertebral fractures and fractures reported by participants where imaging was not performed, was not feasible or where results were inconclusive
Pain assessed by the Brief Pain Inventory (BPI) Short Form measure | Baseline (0), 12 months, 24 months and Final Trial Visit (5 years after baseline)
  Bone pain assessed by the Brief Pain Inventory (BPI) Short Form, a Patient Reported Outcome Measure completed at 4 time-points throughout the trial. The BPI gives two main scores - a pain severity score and a pain interference score. The pain severity score is calculated from the four questions (3-6) about pain intensity. Each item is rated from 0 (no pain) to 10 (pain as bad as you can imagine). The scores from the 4 questions are added together and then divided by 4, giving a severity score out of 10.
  The pain interference score corresponds to Question 9 responses. The seven sub-items are rated from 0 (does not interfere) to 10 (completely interferes). The scores are added together and divided by 7, giving an interference score out of 10.
  Question 2 (pain drawing diagram), Question 7 and Question 8 (pain relief treatment or medication) do not contribute to the scoring.
Quality of life assessed by the SF-36 (v1) Quality of Life | Baseline, 12 months, 24 months and Final Trial Visit (5 years after baseline
  The SF-36 questionnaire consists of 36 generic health questions: 8 health domains of the questionnaire, each of which are summarised (Physical functioning score (10 items), Role-physical score (4 items), Bodily pain (2 items), General health score (5 items), Vitality score (4 items), Social functioning score (2 items), Role-emotional score (3 items), and Mental health score (5 items)). The resulting score for each domain is standardized, to obtain values ranging from 0 to 100, with higher values indicating a better quality of life.Two overall summary measures (physical and mental component scores) are calculated.
Sleep quality assessed by the Pittsburgh Sleep Quality Index (PSQI) measure | Baseline (0), 12 months, 24 months and Final Trial Visit (5 years after baseline)
  Sleep quality as assessed by the Pittsburgh Sleep Quality Index, a Patient Reported Outcome Measure completed at 4 time-points throughout the trial. The Pittsburgh Sleep Quality Index contains 19 self-rated questions. The questions are combined to form seven 'component' scores, each of which has a range of 0-3 points.
  In all cases, a score of 0 indicates no difficulty while a score of 3 indicates severe difficulty. The seven component scores are added to yield one global score, ranging from 0-21 points, 0 indicating no difficulty and 21 indicating severe difficulties in all areas.
Functional status assessed by the Health Assessment Questionnaire (HAQ) measure | Baseline (0), 12 months, 24 months and Final Trial Visit (5 years after baseline)
  The HAQ includes 8 blocks of questions covering difficulties performing simple daily activities. There are 20 questions in total. A 4 point grading system is used to denote degree of difficulty (0=none, 1=some difficulty, 2=great difficulty, 3=not able to perform at all). Each item has a companion aids-devices variable used to record types of assistance the subject uses for his/her usual activities. These variables are coded from 0 to 3 (0 = No assistance is needed, 1 = A special device is used by the subject in his/her usual activities, 2 = The subject usually needs help from another person, 3 = The subject usually needs BOTH a special device AND help from another person). The highest score reported for any component question of the 8 categories determines the score for that category. A global score is calculated by summing the scores for each of the categories and dividing by the number of categories answered.
Adverse events | Through study completion, approximately 5 years
  All adverse events reported throughout the duration of the trial. Summarised by treatment and by severity, causality and seriousness, reporting both the number of events and the number of patients experiencing a given event.
Mechanistic analyses (ITT) | Biological samples collected at Baseline (0), 12 months, 24 months and Final Trial Visit (5 years after baseline)
  Relationship between gender, clinical OI subtype, lowest Bone Mineral Density T score at spine or hip (≤ -2.5 or > -2.5)), type of genetic mutation (mutations of COLIA1 or COLIA2 and biochemical markers of bone turnover with fracture occurrence and response to treatment. Descriptive statistics by treatment group for each subgroup will be presented.
  The primary outcome, defined as the proportion of participants experiencing a clinical fracture validated by x-ray or other imaging, will be analysed for these subgroups. The interaction between subgroup and treatment will be included in the primary and secondary analysis models to determine if the treatment effect differs by subgroup.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Ralston, MD, Principal Investigator — University of Edinburgh
Locations (23):
- St Vincent's Hospital, Dublin, Ireland
- United Kingdom (22):
  - Aberdeen Royal Infirmary, Aberdeen
  - Royal Victoria Hospital, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Bristol Royal Infirmary, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Ninewells Hospital, Dundee
  - Western General Hospital, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow
  - Leicester Royal Infirmary, Leicester
  - Royal Liverpool Hospital and Aintree Hospital, Liverpool
  - Llandough University Hospital, Llandough
  - Guy's and St Thomas' Hospital, London
  - Manchester Royal Infirmary, Manchester
  - James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Nuffield Orthopaedic Centre, Oxford
  - Northern General Hospital, Sheffield
  - University Hospital Southampton, Southampton
  - Royal National Orthopaedic Hospital, Stanmore
  - Haywood Community Hospital, Stoke-on-Trent
  - Wishaw General Hospital, Wishaw

IPD SHARING:
Plan to Share IPD: No
Anonymised aggregate data only will be shared.

REFERENCES:
- See also: Trial webpage — http://edin.ac/topaz-trial

DOCUMENTS (2):
  • Study Protocol (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/37/NCT03735537/Prot_002.pdf
  • Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT03735537/SAP_001.pdf